CLINICAL TRIAL: NCT02139839
Title: A Single-Center Exploratory Study to Evaluate the Effects of the Probiotics L. Rhamnosus GR-1 and L. Reuteri RC-14 on Subjects With Intermediate Nugent Scores
Brief Title: Exploratory Study to Evaluate the Effects of the Probiotics L. Rhamnosus GR-1 and L. Reuteri RC-14
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kimberly-Clark Corporation (Industry)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Western University, Canada (Other); Integrated Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 500-10-0002
Record Dates: First submitted 2014-05-02; First posted 2014-05-15 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Vaginosis, Bacterial
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gelatin pill first (Placebo Comparator)
  Interventions: Other: Lactobacillus capsules; Drug: Placebo gelatin pill
- Lactobacillus capsules first (Experimental)
  Interventions: Other: Lactobacillus capsules; Drug: Placebo gelatin pill

INTERVENTIONS:
Other: Lactobacillus capsules — L. rhamnosus GR-1 and L. reuteri RC-14 capsules manufactured by Chr. Hansen
Drug: Placebo gelatin pill — Placebo Comparator capsules, identical in appearance to the active product; 98% Gelatin with no L. rhamnosus GR-1 and L. reuteri RC- 14.

SUMMARY:
The purpose of this study was to determine whether L. rhamnosus GR-1 and L. reuteri RC-14 delivered via capsules to the vagina of post-menopausal women over a three day course of treatment can restore and maintain a lactobacilli-dominated microbiota. Exploratory analysis of microbial ecology, human microarrays and multiplex immunological assessments are included to characterize potential effects.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read, understand, and sign the Informed Consent Form (ICF);
* Post-menopausal females between the ages of 40 and 80 years old (subjects who have not had a menstrual period for the last 12 months);
* Currently in a mutually monogamous sexual relationship or not sexually active;
* Agree to be sexually abstinent 72 hours prior to each study visit. Also, agree to refrain from intercourse for 48 hours after treatment administration;
* Agree to abstain from the use of any other intravaginal product (e.g. gels, foams, lubricants, douches, etc.) throughout the study period, from the time of screening until Day 47;
* Willing and capable of following all study instructions; and
* Good general health.

Exclusion Criteria:

* Use of vaginal lubricants, or any products applied vaginally within three months prior to Visit 1and throughout the duration of study participation;
* A history or currently undergoing immunosuppressive drug therapy, chemotherapy, or radiation therapy;
* A medical condition which might compromise immune system functions (such as cancer, leucopenia, HIV-positive, or organ transplant);
* Antibiotics and/or antifungal medication use within the last four (4) weeks;
* Oral probiotic supplement use within 3 months prior to Visit 1 and throughout the duration of the study;
* Significant changes in diet during the course of the study based on self-report;
* Induced menopause due to surgical or medical interventions, such as bilateral oophorectomy, hysterectomy, chemotherapy or radiation treatment;
* Currently undergoing local or systemic estrogen therapy who are not willing to alter therapy during the course of the study;
* A Nugent Score of 0 - 3 or greater than 6;
* History of drug or alcohol abuse;
* Currently diagnosed with or being treated for a genital infection or urinary tract infection;
* Individuals with a sexually transmitted disease (self-reported or detected by the Principal Investigator);
* At enrollment, have any social or medical condition, or psychiatric illness that, in the opinion of the Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives;
* Participation in a clinical trial involving an investigational product/device within the past three months; subjects who are scheduled to participate in another clinical study concurrently; and
* Known intolerance or allergy to L. rhamnosus GR-1® or L. reuteri RC-14® or to any product excipients.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline Nugent Score (arbitrary units) after treatment versus Change from baseline Nugent Score after placebo | Baseline Days 15 & 36, post treatment/control Days 19 & 40
  Determine whether L. rhamnosus GR-1 and L. reuteri RC-14 delivered via capsules to the vagina of post-menopausal women over a three day course of treatment can restore and maintain a lactobacilli-dominated microbiota for one week as measured by a decrease in the Nugent Scores from an intermediate score (4 - 6) at baseline to a normal score (0 - 3) following treatment compared to a placebo.

SECONDARY OUTCOMES:
Percent Lactobacilli abundance | Untreated (Days 1, 5, & 15), Baseline Treatment I (Days15), Treatment I (Days 19 & 26), Baseline Treatment II (Day 36), Treatment II (Days 40 & 47)
  Change in lactobacilli abundance before and after probiotic treatment and before and after placebo treatment. Lactobacilli abundance will be calculated as percentage of number of lactobacilli taxon divided by the total number of taxons.
Change in presence of metabolites | Untreated (Days 1, 5, & 15), Baseline Treatment I (Days15), Treatment I (Days 19 & 26), Baseline Treatment II (Day 36), Treatment II (Days 40 & 47)
  Gas chromatography-mass spectrometry will be used to determine changes in metabolites (such as lactate, glutamic acid, and others) before and after probiotic and placebo treatments.
Change in cytokine/chemokine levels | Untreated (Days 1, 5, & 15), Baseline Treatment I (Days15), Treatment I (Days 19 & 26), Baseline Treatment II (Day 36), Treatment II (Days 40 & 47)
  Multiplex ELISA based assay will be used to evaluate the modulation of cytokine and chemokine levels known regulate inflammation and host defense response before and after probiotic and placebo treatment.
Change in global host gene expression | Untreated (Days 1, 5, & 15), Baseline Treatment I (Days15), Treatment I (Days 19 & 26), Baseline Treatment II (Day 36), Treatment II (Days 40 & 47)
  Microarray analysis using GeneChip Human 2.0 ST array will be used to measure gene expression changes (by mRNA analysis) to determine whether there are differences in gene regulation between probiotic, placebo, and no treatment conditions.
Change in self-reported vaginal symptoms | Untreated (Days 1, 5, & 15), Baseline Treatment I (Days15), Treatment I (Days 19 & 26), Baseline Treatment II (Day 36), Treatment II (Days 40 & 47)
  Symptom analysis to evaluate whether probiotic treatment is associated with symptom relief.

CONTACTS AND LOCATIONS:
Locations (1):
- Dorli Herman, London, Ontario, Canada

REFERENCES:
- [Derived] Bisanz JE, Seney S, McMillan A, Vongsa R, Koenig D, Wong L, Dvoracek B, Gloor GB, Sumarah M, Ford B, Herman D, Burton JP, Reid G. A systems biology approach investigating the effect of probiotics on the vaginal microbiome and host responses in a double blind, placebo-controlled clinical trial of post-menopausal women. PLoS One. 2014 Aug 15;9(8):e104511. doi: 10.1371/journal.pone.0104511. eCollection 2014. PMID 25127240